CLINICAL TRIAL: NCT02844985
Title: Genetic Markers in Sexual Addiction
Brief Title: A Study of Gene Polymorphisms Associated With Specific Presentations of Sexual Addiction
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: American Foundation for Addiction Research (Other)
Collaborators: University of Alberta (Other); University of Southern Mississippi (Other)
Responsible Party: Sponsor
Other Study IDs: AFAR 2016-001
Record Dates: First submitted 2016-06-17; First posted 2016-07-26 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Sexual Addiction
Keywords: Sexual Addiction; Genomics; Personality; Polymorphism
MeSH Terms: conditions — Compulsive Sexual Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva specimens will be collected from all participants for genetic evaluation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Addict Group: In-patient and out-patient adult men and women who meet diagnostic criteria for sexual addiction.
  Interventions: Other: No Intervention
- Control Group: Individuals from the general community and college student populations who have no history of identifiable psychopathology.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
The study is intended to identify gene polymorphisms significantly associated with specific behavioral- and preoccupation-typologies of sexual addiction, and to identify additional potential genetic markers of sexual addiction. Research subjects with sexual addiction will be identified from the out-patient and in-patient populations of the investigative sites. Research subjects in the Control Group will be identified from the general population and from the student body of selected colleges. Approximately 1100 subjects will be enrolled in the study. Anticipating 10% drop-out, this is intended to generate a population of approximately 500 men and women clinically diagnosed with sexual addiction, and approximately 500 healthy men and women who do not meet diagnostic criteria for sexual addiction nor have psychopathology who will serve as the control population.

ELIGIBILITY:
Inclusion Criteria:

* Sexual Addict Group

Age >= 18 years

Participating in sexual addiction treatment program

Sexual Addiction Screening Test--Revised (SAST-R) score >= 11

Meets at least 3 diagnostic criteria for sexual addiction

* Control Group

Age >= 18 years

SAST-R score < 6

Exclusion Criteria:

* Sexual Addiction Group

Serious mental illness

Significant cognitive impairment

* Control Group

History of addiction

Current or previous Diagnostic and Statistical Manual (DSM-5) diagnosis

Serious mental illness

Significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sexual Addict Group: individuals undergoing treatment for sexual addiction.
  Control Group: individuals from general community who have no history of addiction or psychopathology
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-08-17 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Gene polymorphisms identified through polymerase chain reaction using fluorescent primers and restriction fragment length polymorphism analysis | Assessed at Enrollment

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Psychological Counseling Services, Scottsdale, Arizona
  - Gentle Path at The Meadows, Wickenburg, Arizona
  - Center for Healthy Sex, Los Angeles, California
  - Triune Therapy Group, Los Angeles, California
  - Pine Grove Behavioral Health and Addiction Services, Hattiesburg, Mississippi
  - Kavod Center, Rochester, New York
  - Center for Healthy Sexuality, Houston, Texas
  - Seattle Christian Counseling, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No